CLINICAL TRIAL: NCT01730196
Title: Fit Body and Soul: A Lifestyle Intervention for Diabetes Prevention Conducted Through African American Churches
Brief Title: Lifestyle Change to Prevent Diabetes Via African-American Churches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Richard Sattin, Professor and Research Director, Department of Emergency Medicine, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R18DK082401 (NIH)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes; Weight Loss
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fit Body and Soul (Experimental): Faith-based adaptation of the Group Life Style Program
  Interventions: Behavioral: Fit Body and Soul
- Wellness education (Active Comparator): A health education program developed from the list of topics provided by the Centers for Disease Control and Prevention (CDC) Guide to Community Prevention Services
  Interventions: Behavioral: Wellness Education

INTERVENTIONS:
Behavioral: Fit Body and Soul
  Arms: Fit Body and Soul
Behavioral: Wellness Education
  Arms: Wellness education

SUMMARY:
Fit Body and Soul is single-blinded, cluster- randomized trial of a faith-based adaptation of the GLB program compared with a health education intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self-described African American
* BMI ≥25kg/m2
* Planning to remain within the community for 1 year
* Non-diabetic

Exclusion Criteria:

* Fasting plasma glucose ≥ 126 mg/dl following at least an 8-hr fast or A1C≥7.0%
* HIV/AIDS
* Active tuberculosis
* Cancer requiring treatment in past 5 years except for cancers that have been cured or in the opinion of the researchers has a good prognosis
* Stroke within the past 6 months
* Cirrhosis of the liver
* Currently pregnant or planning pregnancy within the study period
* Gastric weight-loss surgery
* Weight loss > 10% in past three months for any reason other than childbirth
* Anti-diabetic medications
* Prescription weight- loss medications
* Anti-neoplastic agents
* Anti-psychotic agents that have gluco-corticoid effect
* Oral corticosteroid use >6 weeks
* Unwilling or unable to give informed consent
* Unable to communicate with the church team or research group
* Participation in another research study that would interfere with FBAS

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 604 (Actual)
Dates: Start 2009-09; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Weight change | 12-weeks post intervention

SECONDARY OUTCOMES:
Fasting plasma glucose | 12 week post intervention
physical activity level | 12 week post-intervention
quality of life measures | 12 week post-intervention
cost-effectiveness | 12 week post-intervetnion
  Health Related Quality of Life (HRQoL) which will be assessed using the EQ-5D and the SF-12v2®
hemoglobin A1C | 12 week intervention

OTHER OUTCOMES:
waist circumference | 12 weeks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Sattin, MD, Principal Investigator — Augusta University
Locations (1):
- Georgia Health Sciences University, Augusta, Georgia, United States

REFERENCES:
- [Derived] Rhodes EC, Chandrasekar EK, Patel SA, Narayan KMV, Joshua TV, Williams LB, Marion L, Ali MK. Cost-effectiveness of a faith-based lifestyle intervention for diabetes prevention among African Americans: A within-trial analysis. Diabetes Res Clin Pract. 2018 Dec;146:85-92. doi: 10.1016/j.diabres.2018.09.016. Epub 2018 Sep 28. PMID 30273708
- [Derived] Sattin RW, Williams LB, Dias J, Garvin JT, Marion L, Joshua TV, Kriska A, Kramer MK, Narayan KM. Community Trial of a Faith-Based Lifestyle Intervention to Prevent Diabetes Among African-Americans. J Community Health. 2016 Feb;41(1):87-96. doi: 10.1007/s10900-015-0071-8. PMID 26215167